CLINICAL TRIAL: NCT02731586
Title: Comparative Clinical Evaluation of Osseointegration of Dental Implants Placed With and Without, the Use of Dental Pulp-derived Allogenic Mesenchymal Stem Cells.
Brief Title: Effect on Allogenic Mesenchymal Stem Cells on Osseointegration of Dental Implants
Acronym: MSC&IMPLANTS
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Sri Sai College of Dental Surgery and Research Centre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: SSCDS-IMP-201601
Record Dates: First submitted 2016-04-03; First posted 2016-04-07 (Estimated); Last update posted 2017-10-06 (Actual); Status verified 2017-10

CONDITIONS: Edentulous Alveolar Ridge
Keywords: Dental Implants; Allogenic mesenchymal stem cells; osseointegration; primary stability; resonance frequency analysis; RFA; implants and stem cells; use of stem cells; stem cells

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- osseointegration using Allogenic MSC's (Experimental): Evaluation of Osseointegration of Dental Implants to be done using Allogenic Mesenchymal Stem Cells.Primary and Secondary stability are measured using RFA.
  Interventions: Drug: Allogenic Mesenchymal stem cells

INTERVENTIONS:
Drug: Allogenic Mesenchymal stem cells — Allogenic mesenchymal stem cells are introduced during placement of dental implants.
  Other Names: Transchymal

SUMMARY:
As Regenerative Medicine is the next level in medicinal sciences, the use of mesenchymal cells have become prevalent, Similarly now stem cells are being used in dental research as well in various clinical applications.This study aims to evaluate the overall effect of osseointegration by use of Allogenic Mesenchymal Stem cells while placing dental implants.Healthy subjects will be chosen and dental implants placed bilaterally one with standard surgical protocol and other with the use of Allogenic Mesenchymal Stem cells.The implant stability is checked using Resonance frequency analysis(RFA).The RFA values are statistically evaluated at various intervals and observations will be analysed on both test and control side.

DETAILED DESCRIPTION:
This study prospective single center study . A total of 10 patients are selected to be treated with dental implants for their bilaterally missing edentulous condition, which can be supported by either removable or fixed rehabilitation. The edentulous space can either be in maxilla or mandible. The study is performed at the Department of Implantology (Sri Sai College Of Dental Surgery and Research Center, Vikarabad, India). The study is approved by institutional ethics committee (IEC).

MATERIAL AND METHODS

1. Nobel Biocare Replace Select Dental Implants of size 4.3x10 mm. Healing abutments and implant abutments. 20 Numbers.
2. Nobel Biocare surgical kit
3. Nobel Biocare physio dispenser
4. Transchymal Dental pulp derived Allogenic mesenchymal cells.
5. Ostell ISQ device along with a Smart peg.
6. A Centrifuge.
7. Sterile centrifuge tubes,
8. Sterile pipettes
9. Bone roungers
10. IOPA and KKD Radiographic system
11. Cold saline
12. Suture material and suture needles
13. 70% isopropanol
14. Chiller and a Thermo cool box to carry dry ice
15. Sterile cotton and gauze
16. Mouth mirror
17. Dental examination Probe
18. Needle holder
19. Artery Forceps and scissors.
20. Surgical gown,patient drape, Mouth mask, head cap and surgical gloves
21. High power suction and suction tips.
22. Betadine and chlorhexidine mouthwash.
23. BP blade handle and BP blade no 11,12 and 15
24. Canon DSLR camera
25. Patient models and surgical guide
26. Informed and written consent forms.
27. Case history records
28. Photography and videography waiver consent form
29. Ethical Clearance Certificate
30. CBCT
31. Vital parameters data sheet
32. Diagnostic reports of CBP, RBS, CT, BT and Hg%
33. Antibiotic and anti-allergic prophylaxis.
34. A local anesthetic solution containing 2% lignocaine with 1:100,000-epinephrine and 2ml disposable syringe.
35. Statistical analysis software IBM SPSS version 19.

METHODS

Clinical Procedure

Pre-operative planning is based on clinical and radiographic examination. After thoroughly recording the case history. The following investigations will be done prior to implant placement surgery: CBCT, CBP, CT, BT, Hg%, RBS, Vital signs and other relevant investigations. If all the parameters fulfill the inclusion and exclusion criteria, the patient's impressions are made and study models poured. Intraoral and extraoral photographs are taken. The surgical guide is constructed on the diagnostic models.Stem cells are carried from stem cell bank to the Department of Implantology in a cryovial, safely placed in the special device, which contains dry ice, to maintain the viability of stem cells.

Surgical Procedure

On the day of surgery, the dental operatory is thoroughly fumigated and all the infection control protocols are followed.The participants will be receiving oral and written information about the study and shall be providing the informed consent along with photography and videography waiver consent. Antimicrobial prophylaxis (amoxicillin 1gm) and antihistamine prophylaxis (20mg cetirizine) orally 1 hour before surgery should be given to the patient. The universal precautions protocol is followed to protect yourself, the patients and the dental assistant.The patient is asked to rinse the Oral cavity with chlorhexidine gluconate solution (0.2%) for 1 minute before surgery.

IMPLANT PLACEMENT ON THE CONTROL SIDE

To standardized the protocol the patient's right side is selected as the control side and left side as the test side. The surgical procedure is carried out under local anesthesia containing 2% epinephrine with 1:100,000 epinephrine. The surgical guide is placed on the teeth and is used to mark the position of the implant with round drill till it hits the bone. Mucoperiosteal flaps were raised with mid crestal incision and intrasulcular incision extending to one tooth mesially and other teeth distally. After full thickness flap elevation, the osteotomy sites are prepared using the drilling sequence instructed by the manufacturer.The dental implants Nobel Biocare Replace select (4.3 *10mm size) 4.3mm diameter and 10mm length is selected and placed in the osteotomy site with IF of 40 Ncm.Before approximation of the flap, the primary stability of the implant is recorded with the ostell device, which has a transducer attached to the device and a magnetic attachment smart peg is attached to the implant with a plastic peg holder each implant is measured twice from two different angles,around 90 degrees and parallel to the crestal line.The two measurements buccolingually and mesiodistally are recorded and an average of both the values are taken.The measurements values are then transferred into implant stability quotient (ISQ) units, which are given on a scale of 1- 100, with 100 being the highest degree of stability and it works on the principle of resonance frequency analysis (RFA).The smart peg is removed and Healing abutments are placed over the dental implants. The flap is sutured monofilament sutures 4-0. IOPAR are taken with KKD Radiograph system, which standardizes the distance between the collimator and the IOPAR.

IMPLANT PLACEMENT ON THE TEST SIDE

To standardized the protocol the patient's left side is chosen as the test side.The surgical procedure is carried out under local anesthesia containing 2% epinephrine with 1:100,000 epinephrine. The surgical guide is placed on the teeth and is used to mark the position of the implant with round drill till it hits the bone. Mucoperiosteal flaps were raised with mid crestal incision and intrasulcular incision extending to one tooth mesially and another tooth distally. After full thickness flap elevation, the osteotomy sites are prepared using the drilling sequence instructed by the manufacturer. the stem cells are centrifuged in a sterile environment as per the instructions are given by the stem cell bank.(Thawing protocol )Human mesenchymal stem cells (hMSC) are primary cells which can be successfully used for infusion purpose.The following is the recommended protocol for thawing and infusion of these cells:Remove the Cryovial of stem cells from dry ice,defrost the vial containing stem cells by placing in between both the palms with constant, moderate agitation, until ice in the ampule is no longer visible,immediately disinfect the vial with 70% isopropanol.Working under laminar flow hood, open the vial and transfer the contents to a sterile 15ml centrifuge tube and centrifuge at 3500 RPM for 5 minutes. Decant the supernatant and to the pellet add 1 ml of saline.Mix properly and the cells are ready for infusion at the osteotomy site. Remove the contents in a sterile dappen dish and before infusion of stem cells at the osteotomy site the implant is dipped in the solution for 3 minutes so that the stem cells adhere to the titanium implant surface. The same dental surgeon performs all the cases. The dental implants Nobel Biocare Replace select (4.3 *10mm size) 4.3mm diameter and 10mm length is selected and placed in the osteotomy site with IF of 40 Ncm11.Before approximation of the flap, the primary stability of the implant is recorded with the ostell device, which has a transducer attached to the device and a magnetic attachment smart peg is attached to the implant with a plastic peg holder each implant is measured twice from two different angles,around 90 degrees and parallel to the crestal line.The two measurements buccolingually and mesiodistally are recorded and an average of both the values are taken.The measurements values are then transferred into implant stability quotient (ISQ) units, which are given on a scale of 1- 100, with 100 being the highest degree of stability and it works on the principle of resonance frequency analysis (RFA).The smart peg is removed and Healing abutments are placed over the dental implants. The flap is sutured monofilament sutures 4-0.IOPAR are taken with KKD radiograph system, which standardizes the distance between the collimator and the IOPAR.

POST SURGICAL TREATMENT

The patient is advised to take soft diet for one week and not to spit and rinse for the next 24 hours. Antibiotics, Antihistamines, and NSAIDs must be continued for 3 days. Postoperative edema if any must be controlled with corticosteroids. The sutures are removed one week postoperatively.

Recall visits

Weekly recall of the patient for 12 weeks for evaluation and recording of implant stability measurements with Ostell ISQ device. Patient safety measures are evaluated on every visit like unusual pain, swelling, allergic reaction, inflammation, outgrowth, vital signs, blood assay or any unspecific reactions should be noted down. The emergency contact number is provided to the patient to report any abnormal incidence immediately. The prosthetic part of the treatment is to be carried out after 3 months either with removable or fixed rehabilitation.

Statistical analysis

Descriptive statistics will be computed to summarize the data for its central tendency and dispersion. Two sample t-test will be applied to see the mean change in the outcome variable between experimental and control groups. Repeated measures of ANOVA are being applied to see the time changes between experimental and control groups. Where ever data is not following uniformity, either transforming the data or nonparametric statistical technique will be applied. The analysis will be performed using IBM SPSS Version 19.0.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with bilateral edentulous condition either partial or complete.
2. Patients maintaining adequate oral hygiene
3. Patients with dimensions of alveolar jaw bone in Occlusso-Gingival position >10mm and Bucco-Lingual position < 6mm.

Exclusion Criteria:

1. Systemic diseases which are likely to compromise Implant surgery like Diabetes Mellitus Type I, II and Osteoporosis.
2. Patients with oral parafunctional habits like Bruxism.
3. Smokers who smoke more than 10 cigarettes a day.
4. Self-declared pregnancy or intention to become Pregnant.
5. The use of Regenerative procedures in conjunction with Implant placement.Eg- Grafts ,Sinus Lift procedures.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Determination of Implant Stability with RFA | 3 months
  Dental Implant stability is a measure of primary stability and secondary stability.The Implant stability can be perceived as a combination of Mechanical stability, which is the result of compressed bone holding the implant tightly in place (Primary Stability) and biological stability, which is the result of new bone cells forming at the site of the implant and resultant osseointegration(Secondary stability).The Implant Stability Quotient (ISQ) is a scale of measurement developed by Osstell device for use with the Resonance Frequency Analysis (RFA) method of measuring implant stability. The Implant Stability Quotient is a linear mapping from resonance frequency measured in kHz to the more clinically useful scale of 1-100 ISQ. The higher the ISQ, the more stable is the implant. The Implant stability is measured every fortnight for three months in 10 patients.The values on test side and control side are plotted on the graph and analysed.

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Sufath UR Rehman, (MDS), Principal Investigator — Sri Sai College of Dental Surgery and Research Centre; Venkat Aditya, MDS, Principal Investigator — Sri Sai College of Dental Surgery and Research Centre; Shailaja Reddy, (MDS), Study Director — Sri Sai College of Dental Surgery and Research Centre; Mahendranadh Reddy Kareti, MDS, Study Chair — Sri Sai College of Dental Surgery and Research Centre
Locations (1):
- Sri Sai College Of Dental Surgery and Research Centre, Vikārābād, Telangana State, India

IPD SHARING:
Plan to Share IPD: Undecided
upon total enrollment of participants, it shall be decided.

REFERENCES:
- [Background] Haniffa MA, Collin MP, Buckley CD, Dazzi F. Mesenchymal stem cells: the fibroblasts' new clothes? Haematologica. 2009 Feb;94(2):258-63. doi: 10.3324/haematol.13699. Epub 2008 Dec 23. PMID 19109217
- [Result] Uccelli A, Moretta L, Pistoia V. Mesenchymal stem cells in health and disease. Nat Rev Immunol. 2008 Sep;8(9):726-36. doi: 10.1038/nri2395. PMID 19172693
- [Result] Le Blanc K, Tammik C, Rosendahl K, Zetterberg E, Ringden O. HLA expression and immunologic properties of differentiated and undifferentiated mesenchymal stem cells. Exp Hematol. 2003 Oct;31(10):890-6. doi: 10.1016/s0301-472x(03)00110-3. PMID 14550804
- [Result] Meredith N. Assessment of implant stability as a prognostic determinant. Int J Prosthodont. 1998 Sep-Oct;11(5):491-501. PMID 9922740
- [Result] Lavenus S, Berreur M, Trichet V, Pilet P, Louarn G, Layrolle P. Adhesion and osteogenic differentiation of human mesenchymal stem cells on titanium nanopores. Eur Cell Mater. 2011 Aug 26;22:84-96; discussion 96. doi: 10.22203/ecm.v022a07. PMID 21870339
- [Result] Limet R. [Advantages of side-to-side anastomosis in coronary surgery[(author's transl)]]. Acta Chir Belg. 1976 Jul;75(4):390-401. French. PMID 1087820
- See also: Osseointegration — http://www.osseo.org/
- See also: The Coailation Of Americans For Research Ethics — http://www.stemcellresearch.org/
- See also: Voice of Stemcell Research Community — http://www.isscr.org/
- See also: Stem Cell Research Facts — http://www.stemcellresearchfacts.org/